CLINICAL TRIAL: NCT03764943
Title: Evaluating the Use of Enhanced Recovery Preoperative Immunonutrition and Carbohydrate Loading Strategies in Immediate Autologous and Alloplastic Breast Reconstruction
Brief Title: Immunonutrition and Carbohydrate Loading Strategies in Breast Reconstruction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UW18101; 2018-1107 (Other: Institutional Review Board); A539730 (Other: UW Madison); SMPH/SURGERY/DENTL-PLASTC SRGY (Other: UW Madison); Protocol version 5/8/2020 (Other: HS-IRB UW Madison); NCI-2018-02896 (Other: NCI Trial ID)
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Wound Complication; Wound Heal; Complications Wound; Surgical Wound Infection; Surgical Site Infection; Breast Cancer; Mastectomy; Lymphedema
MeSH Terms: conditions — Surgical Wound Infection; Breast Neoplasms; Lymphedema

STUDY DESIGN:
Intervention Model Description: Prospective cohort study, 2 groups; alloplastic reconstruction and autologous reconstruction, same intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunonutrition Intervention (Experimental): Participants will consume 3 'Impact Advanced Recovery' shakes daily for 5 days prior to surgery 2 hours prior to surgery.
  Interventions: Dietary Supplement: Impact Advanced Recovery

INTERVENTIONS:
Dietary Supplement: Impact Advanced Recovery — immunonutrition shake; nutritional supplement containing amino acids, omega-3 fatty acids, and nucleotides

SUMMARY:
This study is designed to test the following hypothesis: patients undergoing immediate alloplastic and autologous breast reconstruction following mastectomy that receive preoperative immunonutrition will experience a reduction in wound complications in the 30-day postoperative period compared to a standard of care control group (retrospective chart review) of 264 (132 alloplastic + 132 autologous) consecutive breast reconstruction patients prior to 5/25/2018.

DETAILED DESCRIPTION:
Breast reconstruction following mastectomy for breast cancer is one of the most common operations performed by plastic and reconstructive surgeons. Unfortunately, breast reconstruction does not come without complications. Both alloplastic and autologous forms of reconstruction are frequently complicated by wound healing and infectious complications. These complications range from incisional dehiscence requiring prolonged wound care and daily dressing changes, to expander infection and extrusion requiring operative removal, to mastectomy skin flap necrosis so severe that operative debridement is required during a second surgery after declaration of viable skin has occurred.

This study is designed to test the hypothesis that patients undergoing immediate alloplastic and autologous breast reconstruction following mastectomy that receive preoperative immunonutrition will experience a reduction in wound complications in the 30-day postoperative period compared to a standard of care control group (retrospective chart review) of 264 (132 alloplastic + 132 autologous) consecutive breast reconstruction patients prior to 5/25/2018.

The overarching goal of perioperative immunonutrition supplementation is to offset the immune and metabolic dysregulation that occurs in response to surgical stress. The key ingredients that promote this response are amino acids (typically arginine), fatty acids and nucleotides; these can be administered individually but are typically administered together in an enteral or parenteral formula.

The primary outcome measure of the protocol is the incidence of wound complications 30-days post-operative.

Secondary outcome measures are:

1. Rate of return to the operating room in the 30-day postoperative period in patients undergoing immediate alloplastic and autologous breast reconstruction.
2. Average length of stay for patients undergoing autologous reconstruction.
3. Incidence of wound complications and return to the operating room 90-days post-operative throughout expansion process for patients undergoing alloplastic reconstruction.

The study duration will be approximately 33 weeks assuming 100% compliance with the treatment arms in the alloplastic and autologous populations. The time estimate is based on recent trends in operative schedules of 2 immediate alloplastic and 2 immediate autologous breast reconstruction operations weekly with a calculated sample size of 66 patients in each group (total n=132). This sample size was calculated assuming significance level of 0.05, power of 80%, and 50% reduction in wound complications in the treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Medically cleared to undergo oncologic resection and breast reconstructive surgery (including associated anesthesia) at the University of Wisconsin Hospital
* Undergoing unilateral or bilateral immediate alloplastic or autologous breast reconstruction by Drs. Afifi, Garland, Gast, Michelotti, Poore, Rao, or Siebert

Exclusion Criteria:

* Pregnant or breast-feeding women
* Incarcerated women
* Males
* Individuals unable to give consent due to another condition such as impaired decision-making capacity
* Women with intolerance or allergy to any ingredients contained within the Impact Advanced Recovery formula that prevents safe consumption of this product.

  * Impact Advanced Recovery is suitable for lactose intolerance, gluten-free, kosher, and halal diets.
  * We will exclude individuals with galactosemia
* Women who are unable to take oral nutritional supplements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Number of Incidents of Wound Complications 30-days Post-Op | up to 30 days post-op
  Wound complications are defined by the American College of Surgeons National Surgery Quality Improvement Program (ACS-NSQIP) to include surgical site infection (SSI), deep SSI, organ/space SSI, wound disruption/dehiscence, seroma, and skin necrosis.

SECONDARY OUTCOMES:
Number of Patients that Return to the Operating Room 30-days Post-Op | up to 30 days post-op
  The intervention tests the impact of immunonutrition on wound complications post-op. This outcome directly measures this impact by identifying the number of patients that require additional surgery due to wound complications 30-days Post-Op, compared to a retrospective standard of care control group.
Average Length of Hospitalization for Autologous Reconstruction Patients | up to 1 weeks
  The intervention tests the impact of immunonutrition on wound complications post-op. This outcome directly measures this impact by identifying average length of hospitalization for Autologous Reconstruction patients, compared to a retrospective standard of care control group.
Rate of Wound Complications for Alloplastic Reconstruction Patients up to 90-days Post-Op | up to 90 days post-op
  Wound complications are defined by the American College of Surgeons National Surgery Quality Improvement Program (ACS-NSQIP) to include surgical site infection (SSI), deep SSI, organ/space SSI, wound disruption/dehiscence, seroma, and skin necrosis.
Number of Alloplastic Reconstruction Patients that Return to the Operating Room up to 90-days Post-Op | up to 90 days post-op
  The intervention tests the impact of immunonutrition on wound complications post-op. This outcome directly measures this impact by identifying the number of patients undergoing Alloplastic Reconstruction that require additional surgery due to wound complications 90-days Post-Op, compared to a retrospective standard of care control group.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Gast, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/